CLINICAL TRIAL: NCT05617534
Title: A Single-centre, Prospective Case Control Study Evaluating the Impact of a Standardised Aerobic and Strength Exercise Regime on Exercise Capacity, Ventricular Function, and Perceived Quality of Life in Paediatric Fontan Patients
Brief Title: Impact of Exercise Training on Single Ventricle Function in Paediatric Fontan Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Children's Health Ireland (Other Government)
Collaborators: CHI Research & Innovation Office (Unknown)
Responsible Party: Principal Investigator, Adam James, Consultant Paediatric Cardiologist, Children's Health Ireland
Other Study IDs: RSFG-21-ACC13
Record Dates: First submitted 2022-10-24; First posted 2022-11-15 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Univentricular Heart
Keywords: Fontan; Exercise Training; Ventricular Function; Quality of Life
MeSH Terms: conditions — Univentricular Heart

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to learn about how a prescribed Exercise Training Program would affect children living with a Fontan circulation.

From birth, the children who are born with single functioning ventricle will undergo 3-staged Fontan surgery to achieve a unique Fontan circulation, supported by one functioning ventricle. With advancement in surgical technique and medical care, there are increasing number of children living with Fontan circulating surviving into adulthood.

A significant number of these individuals develop complications in their adulthood due to problems related to this unique circulation, including reduced exercise tolerance, heart failure, abnormal heart rhythm or premature death. Many of these children have acquired sedentary lifestyle, and may have lower self-perceived health related quality of life.

Exercise training is a well-established therapy used in adult population with heart failure. It has been shown to be safe in children with congenital heart disease and with Fontan circulation, it improves their aerobic exercise capacity which is associated with better outcomes.

The main question[s] it aims to answer are the impact of a Exercise Training program on:

1. Single ventricle function
2. Exercise capacity
3. Self-perceived quality of life
4. Skeletal muscle mass

Participants will be given a 20-weeks exercise program, 3 sessions of 30 minutes workout weekly, to carry out at home. The following tests will be performed prior to starting and upon completion of the exercise program:

* Echocardiogram
* Cardiopulmonary exercise test
* Body composition scan using a bio-impedance analyser
* Quality of life questionnaires

ELIGIBILITY:
Inclusion Criteria:

* Patients with Fontan circulation, age range 8 to 18 years
* Ability to perform a cardiopulmonary exercise stress test (CPET)
* Free from acute or chronic respiratory illness and/or conditions that might affect exercise performance
* Who have had a Fontan operation at least six months prior.

Exclusion Criteria:

* Existing neuro-disability i.e. with paresis post cerebrovascular accident
* Neurodevelopmental issue with inability to comply with commands.
* Documented life-threatening arrhythmia without implantable cardioverter defibrillator
* Moderate or severe atrio-ventricular valve regurgitation
* Moderate or severe ventricular dysfunction by echocardiography exams
* Acute inflammatory cardiac disease
* documented coronary artery stenosis and/or myocardial ischaemia
* Heart failure requiring hospitalisation in the past year
* Evidence of systemic venous pathway obstruction by echocardiography or catheterisation
* Resting oxygen saturation < 90%
* Systemic ventricular outflow tract stenosis with peak resting systolic gradient > 50mmHg

Ages: 8 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Children aged 8 to 18 years old, who are living with a Fontan circulation, who have met the eligibility criteria listed above.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-01-10 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Single ventricle Function | After a 20 week Exercise training program
  By implementing a prescribed exercise training regime over a 20 week period, a change will be noted in ventricular function at the subclinical state using Echocardiography parameters.

SECONDARY OUTCOMES:
Exercise Capacity | After a 20 week Exercise training program
  By implementing a prescribed exercise training regime over a 20 week period, an improvement will be noted in functional exercise capacity, which will be objectively assessed using cardiopulmonary exercise test.
Self-perceived Quality of life - Generic | After a 20 week Exercise training program
  By implementing a prescribed exercise training regime over a 20 week period, an improvement will be noted in self-reported quality of life, which will be assessed using validated QOL questionnaire - Using Paediatric Quality of Life Inventory, PedsQL v4.0
Self-perceived Quality of life - Cardiac module | After a 20 week Exercise training program
  By implementing a prescribed exercise training regime over a 20 week period, an improvement will be noted in self-reported quality of life, which will be assessed using validated QOL questionnaire - Using PedsQL Cardiac Module v3.0
Skeletal muscle mass | After a 20 week Exercise training program
  By implementing a prescribed exercise training regime over a 20 week period, an improvement will be noted in the skeletal muscle mass, which will be assessed using a non-invasive bio-impedance analyser.

CONTACTS AND LOCATIONS:
Overall Officials: Adam James, MD, Principal Investigator — Children's Health Ireland
Locations (1):
- Children's Health Ireland, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No